CLINICAL TRIAL: NCT05930457
Title: Study of 64Cu-FAPI-XT117 PET/CT in Patients With Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Principal Investigator, Xinlu Wang, chief of nuclear medicine department, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XT-XTR016-1-02
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 64Cu-FAPI-XT117 PET/CT (Experimental)
  Interventions: Drug: 2.5-3.5mCi 64Cu-FAPI-XT117; Drug: 3.5-4.5mCi 64Cu-FAPI-XT117; Drug: 4.5-5.5mCi 64Cu-FAPI-XT117

INTERVENTIONS:
Drug: 2.5-3.5mCi 64Cu-FAPI-XT117 — 64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 2.5-3.5mCi 64Cu-FAPI-XT117 injection.
Drug: 3.5-4.5mCi 64Cu-FAPI-XT117 — 64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 3.5-4.5mCi 64Cu-FAPI-XT117 injection.
Drug: 4.5-5.5mCi 64Cu-FAPI-XT117 — 64Cu-FAPI-XT117 and 18F-FDG PET/CT were performed for each patient(the interval was more than one day and less than four weeks). PET/CT images were acquired 30min, 60min, 120min after 4.5-5.5mCi 64Cu-FAPI-XT117 injection.

SUMMARY:
This is the study of 64Cu-FAPI-XT117, which is an prospective, single-arm phase I clinical study.

ELIGIBILITY:
Inclusion Criteria:

* 1. signed the informed consent
* 2. ≥18 years old
* 3. confirmed as malignant solid tumor by histopathology or clinical judgment
* 4. Patients will undergo 18F-FDG PET/CT examination

Exclusion Criteria:

* 1. Known allergy to components of the investigational drug or its analogues
* 2. suspected to have a certain disease or condition that is not suitable for the study drug
* 3. Known pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 7 days following injection]
  Evaluation of Adverse Events (AE) Using CTCAE

SECONDARY OUTCOMES:
The diagnostic efficacy of 64Cu-FAPI-XT injection in PET/CT imaging of patients with malignant solid tumor | 2 months following injection
  Accuracy (AC), sensitivity (SE), specificity (SP), positive predictive value (PPV)
Change in 'treatment strategy questionnaire' | 2 months following injection
  Referring physicians were asked to complete and return 2 questionnaires. The first assessed the existing treatment plan for the patient without the information from 64Cu-FAPI-XT PET. The second inquired about intended management after receipt of the written clinical report and the 64Cu-FAPI-XT PET images.

OTHER OUTCOMES:
Uptake of the 64Cu-FAPI-XT and optimal scanning specifications for future studies | From first dose of imaging study drug through two hours post dose
Determine impact of administered dose of 64Cu-FAPI-XT on image quality | From first dose of imaging study drug through two hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China